CLINICAL TRIAL: NCT01990937
Title: Effectiveness of Oral Midazolam for Sedation in Patients Undergoing Upper Gastrointestinal Endoscopy
Brief Title: Oral Midazolam for Sedation in Esophagogastroduodenoscopy(EGD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMK-031
Record Dates: First submitted 2013-10-20; First posted 2013-11-25 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Conscious Sedation Failure During Procedure
Keywords: oral midazolam; sedation; premedication; upper gastrointestinal endoscopy; EGD
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral midazolam (Active Comparator): Oral midazolam (5 mg) in 15 mL of apple juice was drunk 30 minutes before EGD
  Interventions: Drug: Oral midazolam
- Apple juice (Placebo Comparator): 15 mL of apple juice was drunk 30 minutes before EGD

INTERVENTIONS:
Drug: Oral midazolam — 5 mg in 15 mL of apple juice, orally 30 minutes before undergoing EGD
  Other Names: Dormicum
  Arms: Oral midazolam

SUMMARY:
Can oral midazolam used for sedation in patients undergoing upper gastrointestinal endoscopy ?

DETAILED DESCRIPTION:
Five mg of midazolam was intake orally about 30 minutes before undergoing perform upper gastrointestinal endoscopy. Declined of anxiety scores was primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective diagnostic EGD
* American Society of Anesthesia (ASA) criteria to be class 1 to 2

Exclusion Criteria:

* History of gastrectomy, esophagectomy, pancreaticoduodenectomy, or other operation on the upper-GI tract
* American Society of Anesthesia (ASA) criteria to be class 3 to 4
* Pregnancy
* Alcoholism
* Drug abuse
* Taking psychotic medications
* Allergy to midazolam.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Difference of Anxiety score | Asked the patient 5 minutes before EGD and then after fully recovery from sedation.
  * Anxiety score is 10-cm scaled visual analog scale.
  * Anxiety score which asked the patient 5 minutes before EGD, called "Pre EGD anxiety score"
  * Anxiety score which asked the patient after fully recovery, called "During EGD anxiety score".
  * Difference of anxiety score means "Pre EGD minus During anxiety score".
  * Fully recovery means fully gain of consiouness (time, place, person).

SECONDARY OUTCOMES:
Overall tolerance | Asked the patient after fully recovery from sedation.
  Fully recovery means fully gain of consiouness (time, place, person).
  Overall tolerance was grading into 4 levels;
  * Poor : Very uncomfortable during the entire procedure
  * Fair : Uncomfortable during most of the procedure
  * Good : Believes the procedure was generally comfortable, there were portions of procedure during which sedation could have been given
  * Excellent : Believes the procedure was comfortable, no additional sedation was needed

OTHER OUTCOMES:
Amnesia score | Asked the patient after fully recovery from sedation.
  Fully recovery means fully gain of consiouness (time, place, person).
  Amnesia score was grading into 4 levels;
  1. = Patient unable to recall any portion of procedure
  2. = Able to recall and describe some portion of procedure
  3. = Able to recall and describe most of procedure
  4. = Able to recall and describe entire procedure
Overall satisfaction | Asked the patient after fully recovery from sedation.
  Fully recovery means fully gain of consiouness (time, place, person). Overall satifaction was 10-cm scaled visual analog scale.
Willing to repeat EGD | Asked the patient after fully recovery from sedation.
  Fully recovery means fully gain of consiouness (time, place, person). Willing to repeat EGD was defined to "Yes or No".
Vital signs | Vital signs were measured at 5 minutes before EGD then measured every 5 minutes during EGD until the patient was fully recovery after the EGD was finished.
  Vital signs were blood pressure(mmHg), heart rates(beats per minute), respiratory rates(per minute) and oxygen saturation(percents).

CONTACTS AND LOCATIONS:
Overall Officials: Chaipichit Puttapitakpong, Doctor, Principal Investigator — Division of gastroentrology, Department of Medicine, Phramongkutklao hospital
Locations (1):
- Division of Gastroenterology, Department of Medicine, Phramongkutklao hospital, Bangkok, Thailand